CLINICAL TRIAL: NCT05391984
Title: Effects of Activity Versus Structural Oriented Treatment Approach on Pain, Range of Motion, and Function in Patients With Frozen Shoulder.
Brief Title: Effects of Activity Versus Structural Oriented Treatment Approach in Patients With Frozen Shoulder.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0118
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Frozen Shoulder
Keywords: frozen shoulder; manual therapy; proprioceptive neuromuscular facilitation; neuroplasticity; diabetes
MeSH Terms: conditions — Bursitis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity oriented (Experimental): Activity-oriented therapy will be given to 15 patients which will train the structures around the shoulder in different activities of daily life.
  Interventions: Other: Activity oriented treatment
- Structural oriented (Experimental): Structural-oriented therapy will be given to 15 patients including a fixed sequence of physiotherapy techniques.
  Interventions: Other: Structural oriented treatment

INTERVENTIONS:
Other: Activity oriented treatment — 15 patients will be treated with activity oriented therapy. All subjects will receive 20 therapeutic sessions, 5 times a week over the time span of 4 weeks.
  Arms: Activity oriented
Other: Structural oriented treatment — 15 patients will be treated with structural oriented therapy. All subjects will receive 20 therapeutic sessions, 5 times a week over the time span of 4 weeks.
  Arms: Structural oriented

SUMMARY:
The aim of this study is to compare the effects of activity versus structural oriented treatment approach on pain, range of motion, and function in diabetic patients with frozen shoulder.

DETAILED DESCRIPTION:
Frozen shoulder, also known as adhesive capsulitis, is a condition of uncertain etiology, characterized by shoulder stiffness, severe pain, significant restriction of range of motions, and limitation in participation in socio-economical life. According to a concept, pain causes changes in the brain making it learn the non-use, and therefore, even after healing of peripheral structures has occurred, the brain may not be able to organize voluntary actions owing to the induced central changes. Physical therapy plays an important role to bring pain relief and return of functional motion in frozen shoulder and there are many approaches available that can be used but literature on treatments based on neuroplasticity is comparatively less.

According to the research available, neuroplasticity has been effective in treating frozen shoulder. Similarly, PNF, home exercises, and joint mobilizations have also proven to be effective. The effects of the activity related and structural-oriented treatment on the frozen shoulder has not been addressed in diabetic patients yet. More RCTs are required to determine the best treatment for managing adhesive capsulitis in diabetics. Therefore, this research will be conducted which will compare the activity-based approach and the conventional approach to treating frozen shoulder in diabetics. The results may open new aspects of treating frozen shoulder in diabetics which can be cost-effective as well.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with frozen shoulder, limited ROM, and pain in the shoulder region
* Patients with diabetes from 10+ years

Exclusion Criteria:

* History of headaches and dizziness
* Pain and limited ROM in the cervical spine
* Pain and limited ROM in temporomandibular joint

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NPRS for pain | 4th week
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Goniometer for range of motion | 4th week
  It will be used to measure flexion, extension, abduction, adduction, and internal and external rotation of shoulder.
SPADI for pain and disability | 4th week
  Shoulder pain and disability index include thirteen questions measuring pain and disability on an eleven-point scale. O being no pain, difficulty and 10 being worst pain and difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman Bashir, PhD, Principal Investigator — Riphah International University
Locations (1):
- Social security hospital, Kot Lakhpat, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lho YM, Ha E, Cho CH, Song KS, Min BW, Bae KC, Lee KJ, Hwang I, Park HB. Inflammatory cytokines are overexpressed in the subacromial bursa of frozen shoulder. J Shoulder Elbow Surg. 2013 May;22(5):666-72. doi: 10.1016/j.jse.2012.06.014. Epub 2012 Sep 21. PMID 22999851
- [Background] Cho CH, Lee YH, Kim DH, Lim YJ, Baek CS, Kim DH. Definition, Diagnosis, Treatment, and Prognosis of Frozen Shoulder: A Consensus Survey of Shoulder Specialists. Clin Orthop Surg. 2020 Mar;12(1):60-67. doi: 10.4055/cios.2020.12.1.60. Epub 2020 Feb 13. PMID 32117540
- [Background] Cho CH, Bae KC, Kim DH. Treatment Strategy for Frozen Shoulder. Clin Orthop Surg. 2019 Sep;11(3):249-257. doi: 10.4055/cios.2019.11.3.249. Epub 2019 Aug 12. PMID 31475043
- [Background] Abrassart S, Kolo F, Piotton S, Chih-Hao Chiu J, Stirling P, Hoffmeyer P, Ladermann A. 'Frozen shoulder' is ill-defined. How can it be described better? EFORT Open Rev. 2020 May 1;5(5):273-279. doi: 10.1302/2058-5241.5.190032. eCollection 2020 May. PMID 32509332
- [Background] Klug S, Anderer P, Saletu-Zyhlarz G, Freidl M, Saletu B, Prause W, Aigner M. Dysfunctional pain modulation in somatoform pain disorder patients. Eur Arch Psychiatry Clin Neurosci. 2011 Jun;261(4):267-75. doi: 10.1007/s00406-010-0148-4. Epub 2010 Oct 6. PMID 20924589
- [Background] Vartiainen N, Kirveskari E, Kallio-Laine K, Kalso E, Forss N. Cortical reorganization in primary somatosensory cortex in patients with unilateral chronic pain. J Pain. 2009 Aug;10(8):854-9. doi: 10.1016/j.jpain.2009.02.006. PMID 19638329
- [Background] Horst R, Maicki T, Trabka R, Albrecht S, Schmidt K, Metel S, von Piekartz H. Activity- vs. structural-oriented treatment approach for frozen shoulder: a randomized controlled trial. Clin Rehabil. 2017 May;31(5):686-695. doi: 10.1177/0269215516687613. Epub 2017 Jan 13. PMID 28081633
- [Background] Saab CY. Pain-related changes in the brain: diagnostic and therapeutic potentials. Trends Neurosci. 2012 Oct;35(10):629-37. doi: 10.1016/j.tins.2012.06.002. Epub 2012 Jul 3. PMID 22763295
- [Background] Tedla JS, Sangadala DR. Proprioceptive neuromuscular facilitation techniques in adhesive capsulitis: a systematic review and meta-analysis. J Musculoskelet Neuronal Interact. 2019 Dec 1;19(4):482-491. PMID 31789299
- [Background] AN Y, PARK C. EFFECTS OF A DEEP LEARNING-BASED SMARTPHONE APPLICATION ON SHOULDER ABDUCTION KINEMATICS AND BRAIN ACTIVATION IN ADHESIVE CAPSULITIS: A RANDOMIZED CONTROLLED TRIAL. Journal of Mechanics in Medicine and Biology. 2021:2140076.